CLINICAL TRIAL: NCT07329309
Title: The Effect of Post-Caesarean Section Pranayama Breathing Exercises on Pain and Postpartum Comfort: A Randomised Controlled Trial
Brief Title: Post-Caesarean Pranayama and Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: KTO Karatay University (Other)
Responsible Party: Principal Investigator, Hafize Dağ Tüzmen, Asst.Prof., KTO Karatay University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Pranayama
Record Dates: First submitted 2025-12-12; First posted 2026-01-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Postoperative Pain
Keywords: caesarean section; pain; pranayama; comfort
MeSH Terms: conditions — Pain, Postoperative; Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pranayama group (Experimental)
  Interventions: Behavioral: pranayama breathing exercises
- control group (No Intervention)

INTERVENTIONS:
Behavioral: pranayama breathing exercises — In this study, a pranayama breathing exercise protocol lasting approximately 14-15 minutes will be applied, aiming to increase relaxation and physiological well-being. Participants will prepare for the exercise in a supported and comfortable sitting position, breathing through the nose. The protocol consists of 3 minutes of diaphragmatic breathing, 5 minutes of alternate nostril breathing (Nadī Shodhana), 3 minutes of Ujjayi breathing, and 3 minutes of long, slow exhalation techniques. The exercises will be conducted with one-on-one guidance by a trained researcher; participants' comfort and any signs of discomfort will be monitored, and the exercise will be terminated if necessary.
  Arms: Pranayama group

SUMMARY:
This study aims to investigate the effect of pranayama breathing exercises on postoperative pain and postpartum comfort levels in women following caesarean section, with the objective of providing important evidence for the integration of non-pharmacological methods into postpartum care.

ELIGIBILITY:
Inclusion Criteria:

* Undergone a caesarean section under spinal anaesthesia
* Reported a post-operative pain level of at least 4 on the Numerical Rating Scale (NRS)
* Knowledge of Turkish
* Ability to communicate effectively with the research team
* Volunteer to participate in the study and provide written consent

Exclusion Criteria:

* Having given birth by emergency caesarean section
* Presence of pregnancy complications (e.g. pre-eclampsia, gestational diabetes, placenta praevia)
* History of chronic pain or analgesic dependence
* Requirement for admission to the intensive care unit in the early postoperative period
* Need for additional surgical intervention
* Development of significant intraoperative or postoperative complications
* Refusal to exercise or intolerance to exercise
* Failure to comply with study procedures
* Withdrawal of consent
* Incomplete follow-up
* Development of a new medical condition during the study that could affect the results

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Postpartum period- ceserian section
Enrollment: 100 (Estimated)
Dates: Start 2026-02-05 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-04-13 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Post-Cesarean Postoperative Pain Intensity | Pain assessments will be repeated at 6, 12, 24 hours postoperatively in both groups.
  Postoperative pain intensity will be assessed using the Visual Analog Scale (VAS), a 10-cm horizontal line where 0 indicates "no pain" and 10 indicates "worst imaginable/unbearable pain." Higher scores indicate greater pain severity.
  Pain scores will be recorded at baseline (preoperative) and at predefined postoperative time points. The outcome measure is defined as the change in VAS pain score from baseline.Pain will be assessed with a 10 cm visual analog scale "0" means no pain and "10" means unbearable pain. The assessment will be done before and at the end of the study.

SECONDARY OUTCOMES:
Postnatal Comfort Level | Comfort assessments will be repeated at 6, 12, 24 hours postoperatively in both groups.
  Postnatal comfort will be assessed using the Postnatal Comfort Survey, a validated instrument designed to evaluate physical, psychospiritual, sociocultural, and environmental comfort in the postpartum period.
  Higher scores indicate greater postnatal comfort. Accordingly, the lowest score that can be obtained on the scale is 34, and the highest score is 170.

CONTACTS AND LOCATIONS:
Locations (1):
- Kto Karatay University, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No